CLINICAL TRIAL: NCT00557180
Title: Obesity, Inflammation and Response to Therapy in Asthma - Ancillary to Asthma Clinical Research Network (ACRN) Trials
Brief Title: Examining the Link Between Obesity, Inflammation, and Response to Asthma Medications
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1423; R01HL090982 (NIH)
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Asthma; Obesity
Keywords: Steroid Resistance; Inflammation
MeSH Terms: conditions — Asthma; Obesity; Inflammation | interventions — Beclomethasone; Tiotropium Bromide; Salmeterol Xinafoate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BASALT: Participants in the ACRN BASALT study
  Interventions: Drug: Beclomethasone dipropionate HFA
- TALC: Participants in the ACRN TALC study
  Interventions: Drug: Tiotropium bromide; Drug: Salmeterol xinafoate

INTERVENTIONS:
Drug: Beclomethasone dipropionate HFA — Participants will receive the BASALT and TALC study drugs as determined in those protocols NCT00495157, NCT00565266. This study is ancillary to those trials and observational only and does not have any control over study drug allocation
  Other Names: QVAR® 40 mcg or QVAR® 80 mcg
  Groups: BASALT
Drug: Tiotropium bromide — Participants will receive the BASALT and TALC study drugs as determined in those protocols NCT00495157, NCT00565266. This study is ancillary to those trials and observational only and does not have any control over study drug allocation
  Other Names: Spiriva®
  Groups: TALC
Drug: Salmeterol xinafoate — Participants will receive the BASALT and TALC study drugs as determined in those protocols NCT00495157, NCT00565266. This study is ancillary to those trials and observational only and does not have any control over study drug allocation
  Other Names: Serevent®
  Groups: TALC

SUMMARY:
Asthma is a common, long-term disease that is caused by inflammation of the airways. Inflammation also plays a role in obesity and may affect the way a person responds to asthma medication. This study will examine the relationship between obesity and inflammation and the effect they have on response to corticosteroid asthma medications.

DETAILED DESCRIPTION:
Asthma affects 20 million people in the United States. It can be caused by many factors, including exposure to tobacco smoke, infections, and other allergens. Recent research suggests that there may be a relationship between obesity and asthma. It is not fully understood how these two conditions are linked, but inflammation may play a role. Obesity-related inflammation may increase the risk of airway inflammation, thereby elevating the risk of developing asthma. Increased inflammation related to obesity may also reduce the effectiveness of inhaled steroid asthma medications, including glucocorticoids. Compared with people of normal weight, people who are overweight or obese may have a higher risk of developing glucocorticoid insensitivity, resulting in intolerance to glucocorticoid medications. The purpose of this study is to examine the effect that obesity has on glucocorticoid insensitivity and inflammation. This study will also examine differences in the response to asthma steroid medications between people who are overweight or obese and those who are not.

This study will use previously collected data from participants in two clinical trials of the NHLBI-funded Asthma Clinical Research Network (ACRN): the Best Adjustment Strategy for Asthma in Long Term (BASALT) study (NCT00495157) and the Tiotropium Bromide as an Alternative to Increased Inhaled Corticosteroid in Patients Inadequately Controlled on a Lower Dose of Inhaled Corticosteroid (TALC) study. There will be no additional study visits specifically for this study. Researchers will examine blood samples collected at participants' first BASALT or TALC study visit to analyze levels of inflammation biomarkers (including tumor necrosis factor-alpha [TNF-α], interleukin-6 [IL-6], and leptin) and proinflammatory cytokines levels, which influence glucocorticoid insensitivity. Additional BASALT and TALC study data, including lung function, asthma symptoms, and asthma exacerbations, will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Participation in either the BASALT or TALC studies of the Asthma Clinical Research Network. Inclusion and exclusion criteria are as determined by those studies, NCT00495157, NCT00565266.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the BASALT and TALC studies. Participants will receive the BASALT and TALC study drugs as determined in those protocols NCT00495157, NCT00565266. This study is ancilary to those trials and observational only and does not have any control over study drug allocation
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Measures of lung function; asthma symptoms and exacerbations; quality of life; rescue medication usage; inflammation and oxidative stress biomarkers; and the effect these factors have on glucocorticoid insensitivity | Measured at Week 36 for BASALT participants and Week 46 for TALC participants

CONTACTS AND LOCATIONS:
Overall Officials: E. R. Sutherland, MD, MPH, Principal Investigator — National Jewish Medical & Research Center
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Sutherland ER, Goleva E, Jackson LP, Stevens AD, Leung DY. Vitamin D levels, lung function, and steroid response in adult asthma. Am J Respir Crit Care Med. 2010 Apr 1;181(7):699-704. doi: 10.1164/rccm.200911-1710OC. Epub 2010 Jan 14. PMID 20075384
- See also: Click here for the Asthma Clinical Research Network (ACRN) Web site. — http://www.acrn.org